CLINICAL TRIAL: NCT02861885
Title: Detection and Characterization of Sessile Serrated Lesions (SSL) of the Right Colon
Acronym: Lesion SSL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0158
Record Dates: First submitted 2016-08-02; First posted 2016-08-10 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Neoplasm; Sessile Serrated Lesion; Neoplasms
Keywords: Colonoscopy; sessile serrated lesions; chromoendoscopy; narrow band imaging; Indigo Carmin®; Pit pattern; Kudo classification; NICE classification; neoplasms by histologic type
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms; Neoplasms by Histologic Type

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lesion SSL: Patient cohort referred by colonoscopy screening indication, digestive syndrome or monitoring, with ascendant colon macroscopic SSL suspicion throughout white light during colonoscopy
  Interventions: Other: Chromoendoscopy

INTERVENTIONS:
Other: Chromoendoscopy — Colonoscopy will run in accordance with standard procedure, including air insufflation throughout the endoscope rise. The endoscope will be a Olympus NBI videoscope (180 series and latest). First, progression will run until caecum without systematic terminal ileum intubation. Polyps will be searched out during descent phase. The patient will be eligible as soon as the operator suspects an ascendant colon SSL with white light. The operator will have to initiate the WLI colonoscopy. If a SSL is suspected in the colon, the operator will run at the same time, a NBI colon examination, then an indigo carmine chromoendoscopy colon examination. Each lesion will be pictured before and after mucus clean-up. Lesions biopsy or resection will be ran in accordance with standard procedure.

SUMMARY:
There are a few studies regarding Sessile Serrated Lesions (SSL). They are recently identified as precancerous lesions. Yet, digestive tract serrated lesions would be part of a new colic carcinogenesis way : the serrated tumor way. Evolution from polyp to cancer would be faster than through the usual adenoma to cancer way. It would be then responsible of a lot of "missed" lesions or interval cancer. The missed SSL rate is estimated at between 27% and 59%.

Current diagnosis methods show weakness to identify those SSL. In order to improve their detection, the investigators dispose of several coloration techniques. Indigo carmine chromoendoscopy enhance neoplastic lesion detection as part of the hereditary rectal carcinoma screening. NBI electronic coloration, which is faster and easier has not shown any efficacy on the adenoma detection rate, except for patients with Lynch syndrome.

The objective is to better describe the SSL endoscopic semiology (detection and characterization) and to establish standards for the endoscopic techniques in order to improve the colonoscopy diagnosis quality. The investigators propose to evaluate 2 fundamental endoscopic techniques (Narrow Band Imaging (NBI) and indigo carmine), widely used for other indications, in comparison with the White Light technique (WLI).

Therefore, the investigators propose a prospective, observational, multicentric cohort study in order to 1) define SSL endoscopic various aspects 2) establish which technique (white light, Narrow Band Imaging, indigo carmine chromoendoscopy) is the best to diagnose SSL, namely detection and characterization 3) evaluate the multifocal dimension rate for those lesions at ascending colon level.

The diagnosis impact is immediate, and could allow to consider an update for boh endoscopic NICE and Kudo Pit Pattern classification, and good practice guidances for colonoscopic diagnosis. Better SSL detectability thus their systematic resection could have a long term effect in reducing both colon cancer rate and interval cancer

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Patient having an indication for colonoscopy to detect colorectal neoplastic lesions, which meet at least one of the following conditions :
* Positive fecal occult blood test
* 1st degree family history of colorectal cancer or adenoma before 60 years of age
* Personal history of colorectal adenoma or colorectal cancer
* Unexplained digestive symptoms after 50 years of age or those not responding to symptomatic treatment : modification of bowel movements, abdominal pains
* Isolated or repeated rectal bleeding after 50 years of age or occult bleeding
* Acromegaly
* Infectious endocarditis with digestive bacteria
* Suspicion of sessile serrated lesion in the right colon
* None opposite of patient for participating

Exclusion Criteria:

* History of digestive resection as resection of the right colon (right ileocolectomy, right hemicolectomy) or large colic resection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population being studied is the cohort of patients referred for a colonoscopy resulting screening indication, digestive syndrome or monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2022-04-24 (Estimated); Study Completion 2022-04-24 (Estimated)

PRIMARY OUTCOMES:
patients with sessile serrated lesions | at colonoscopy day (Day 1)
  Proportion of patient for whom at least one new SSL has been shown macroscopically through NBI and/or indigo carmine chromoendoscopy but not detected with WLI

SECONDARY OUTCOMES:
PARIS classification | at colonoscopy day (Day 1)
  All SSL will be characterized using the PARIS classification of colorectal polyps
Kudo's pit pattern classification | at colonoscopy day (Day 1)
  All SSL will be characterized using the Kudo's pit pattern classification for colorectal neoplasms
NICE classification | at colonoscopy day (Day 1)
  All SSL will be characterized using the Narrow band imaging International Colorectal Endoscopic (NICE) of small colorectal polyps.
Specific mean of macroscopically detected SSL | at colonoscopy day (Day 1)
  Comparison of the mean number of SSL per technique (white light, Narrow Band Imaging, indigo carmine chromoendoscopy)
SSL histologic characterization | histopathological results (up to 2 weeks)
  All SSL will be characterized using the Vienna classification of gastrointestinal epithelial neoplasia
False positive | histopathological results (up to 2 weeks)
  Number of suspected SSL macroscopically but unconfirmed histologically
False negative | histopathological results (up to 2 weeks)
  Number of polyps not identified as SSL, but reclassified by histological results
Detection techniques diagnosis performance | at colonoscopy day (Day 1)
  Proportion of macroscopically suspected SSL by one of the 3 techniques (white light, Narrow Band Imaging, indigo carmine chromoendoscopy) and confirmed by centralized review (macro true positive)
Detection techniques diagnosis performance | at colonoscopy day (Day 1)
  Proportion of macroscopically suspected SSL by one of the 3 techniques (white light, Narrow Band Imaging, indigo carmine chromoendoscopy) but not confirmed by centralized review (macro false positive)
Detection techniques diagnosis performance | at colonoscopy day (Day 1)
  Proportion of macroscopically not suspected SSL by one of the 3 techniques (white light, Narrow Band Imaging, indigo carmine chromoendoscopy) and yet seen by centralized review (macro false negative)
Detection techniques diagnosis performance | at colonoscopy day (Day 1)
  Proportion of macroscopically suspected SSL by one of the 3 techniques (white light, Narrow Band Imaging, indigo carmine chromoendoscopy) and confirmed by expert center (true positive)
Detection techniques diagnosis performance | at colonoscopy day (Day 1)
  Proportion of macroscopically suspected SSL by one of the 3 techniques (white light, Narrow Band Imaging, indigo carmine chromoendoscopy) but not confirmed by centralized review (false positive)
Detection techniques diagnosis performance | at colonoscopy day (Day 1) + histopathological results (up to 2 weeks)
  Proportion of macroscopically suspected SSL by the endoscopist and confirmed as SSL with histological results from expert center (false negative)

CONTACTS AND LOCATIONS:
Overall Officials: Christine CHAMBON-AUGOYARD, MD, Principal Investigator — Hospices Civils de Lyon, Hôpital E Herriot, Service d'hépatogastroentérologie, 5 place d'Arsonval, 69437 LYON cedex 03, France
Locations (6):
- France (6):
  - Hôpital Estaing, CHU Clermont Ferrand, NHE Service d'Hépato-gastroentérologie, 1 place Lucie Aubrac, Clermont-Ferrand
  - Centre Hospitalier Saint JOSEPH Saint Luc, Service d'hépato-gastroentérologie, 20 quai Claude Bernard, Lyon
  - Hospices Civils de Lyon, Hôpital de la Croix Rousse, Service d'hépato-gastroentérologie, 103 Grande-Rue de la Croix Rousse, Lyon
  - Hospices Civils de Lyon, Hôpital E Herriot, Service d'hépatogastroentérologie, 5 place d'Arsonval, Lyon
  - Hospices Civils de Lyon, Hôpital Lyon Sud, Service d'hépato-gastroentérologie, Chemin Grand Revoyet, Pierre-Bénite
  - Centre Hospitalier Villefranche sur Saône, Service d'Hépato-gastroentérologie, Plateux d'Ouilly Gleize, Villefranche-sur-Saône